CLINICAL TRIAL: NCT06349772
Title: Zynrelef vs Exparel: The Battle of Postoperative Pain Control After Robotic Sleeve Gastrectomy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FY2024-203
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Post Operative Pain
Keywords: robotic surgery; sleeve gastrectomy; zynrelef; exparel
MeSH Terms: conditions — Pain, Postoperative | interventions — bupivacaine-meloxicam drug combination

STUDY DESIGN:
Intervention Model Description: randomizing study participants to either Exparel or Zynrelef at the closure site of robotic sleeve gastrectomy and assessing their pain control postoperatively
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Patients who receive zynrelef (Experimental): Those who get zynrelef injected at the at the 12mm port incision
  Interventions: Drug: Zynrelef
- Patients who receive exparel (Experimental): those who get exparel injected at the 12mm port incision
  Interventions: Drug: Exparel

INTERVENTIONS:
Drug: Zynrelef — Zynrelef will be injected at the 12mm port site
  Arms: Patients who receive zynrelef
Drug: Exparel — Exparel will be injected at the 12mm port site
  Arms: Patients who receive exparel

SUMMARY:
The purpose of this study is to evaluate the use of an injectable combination of bupivacaine and meloxicam (Zynrelef) vs injectable liposomal bupivacaine (Exparel), two extended local anesthesia strategies currently approved by FDA and on the market for post-surgical pain control. The investigators plan on randomizing study participants to either Exparel or Zynrelef at the closure site of robotic sleeve gastrectomy and assessing their pain control postoperatively both in the hospital and at home. The investigators will measure the outcome of two drugs, Zynrelief, and Exparel on postoperative pain score -using the NRS pin score up to 72 hours after surgery. The total opioid use will be recorded in forms that will be used to measure pain score and total opioid use and will be collected to the Excel sheet. The cost of the drug will be calculated for internal use for Hospital purpose only.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-65 years old
2. Scheduled or being scheduled to undergo robotic sleeve gastrectomy by Dr. Goyal.
3. Is able to provide written informed consent.
4. Is able to adhere to the study visit schedule and complete all study assessments.

Exclusion Criteria:

1. Positive urine drug screen prior to surgery
2. History of substance abuse in the past year-by self report
3. Patient with ongoing daily narcotic use at the time of surgery-by self report
4. Inability to understand informed consent or read English/Spanish
5. Pregnant or lactating patients
6. Prisoners
7. Patients with renal or hepatic failure
8. Bupivacaine use within 96 hours of operation
9. Patient intolerant of opiates, nonsteroidal anti-inflammatory drug s, acetaminophen, or Zynrelef and Exparel. Subjects in all cohorts must not have any contraindications to any of the protocol-specified drugs
10. Patient with a history of asthma, urticaria, or other allergic-type reactions after taking aspirin or other NSAIDs. Severe, sometimes fatal, anaphylactic reactions to NSAIDs have been reported in such patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain score | 72 hours
  this will be measured using a numerical rating scale. The scale is 0-10 with 0 being no pain and 10 being the worst pain of their life

SECONDARY OUTCOMES:
Total postoperative opioid use | 72 hours
  total amount of pain medications used postoperatively converted into morphine equivalents
Proportion of total rescue medication use | 72 hours
  the amount of times a rescue medication had to be used

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Other researchers will be involved with gathering and interpreting data
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: one year
Access Criteria: Access will be given through the EMR